CLINICAL TRIAL: NCT05741853
Title: Cognitive Reserve and Linguistic Resilience in Bilingual Hispanics With Primary Progressive Aphasia
Brief Title: Cognitive Reserve and Response to Speech-Language Intervention in Bilingual Speakers With Primary Progressive Aphasia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01AG080470 (NIH)
Record Dates: First submitted 2023-02-03; First posted 2023-02-23 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Primary Progressive Aphasia; Dementia; Dementia, Frontotemporal; Alzheimer Disease; Neurodegenerative Diseases; Frontotemporal Lobar Degeneration; Apraxia, Motor; Dysarthria; Communication Disorders; Language Disorders; Speech Disorders; Neurocognitive Disorders; Aphasia; Bilingual Aphasia
Keywords: Dementia, ADRD; Bilingualism; Multilingualism; Primary Progressive Aphasia; Bilingual Primary Progressive Aphasia; Cognitive Reserve; Language Decline; Bilingual Language Decline; Speech-Language Therapy; Bilingual Speech-Language Therapy; Spanish speakers; Spanish-Catalan Bilinguals; Spanish-English Bilinguals; Hispanic; Catalán; Catalan; Spanish; Castellano; Speech Therapy; Latino; Cognition
MeSH Terms: conditions — Aphasia, Primary Progressive; Dementia; Frontotemporal Dementia; Alzheimer Disease; Neurodegenerative Diseases; Frontotemporal Lobar Degeneration; Apraxias; Dysarthria; Communication Disorders; Language Disorders; Speech Disorders; Neurocognitive Disorders; Aphasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lexical Retrieval Training (Experimental): Naming intervention for individuals with logopenic or semantic variant PPA.
  Interventions: Behavioral: Video-Implemented Script Training for Aphasia (VISTA); Behavioral: Lexical Retrieval Training (LRT)
- Video Implemented Script Training for Aphasia (Experimental): Script training intervention for individuals with nonfluent/agrammatic PPA.
  Interventions: Behavioral: Video-Implemented Script Training for Aphasia (VISTA); Behavioral: Lexical Retrieval Training (LRT)

INTERVENTIONS:
Behavioral: Video-Implemented Script Training for Aphasia (VISTA) — Participants with nonfluent/agrammatic variant primary progressive aphasia (PPA) or a predominantly nonfluent profile work on producing personally relevant scripts of 4-6 sentences in length. Length and complexity of scripts are individually tailored. The participant completes two (one hour each) teletherapy sessions per week with a clinician targeting clear and accurate script production, script memorization, and conversational usage of scripts. The participant completes 30 minutes of independent, computer-based practice 5-7 times per week, during which they speak in unison with a video/audio model of a healthy speaker clearly articulating the scripts.
  Other Names: Script training
Behavioral: Lexical Retrieval Training (LRT) — Participants with logopenic variant PPA, participants with semantic variant PPA, and participants with a predominantly anomic profile will work on producing spoken and written names of personally relevant target items using a self-cueing hierarchy. Treatment focuses on the use of strategies that capitalize on spared cognitive-linguistic abilities to support word retrieval. The participant completes two (one hour each) teletherapy sessions per week with a clinician plus 30 minutes of additional independent, computer-based practice exercises 5-7 times per week.
  Other Names: Naming intervention

SUMMARY:
Difficulties with speech and language are the first and most notable symptoms of primary progressive aphasia (PPA). While there is evidence that demonstrates positive effects of speech-language treatment for individuals with PPA who only speak one language (monolinguals), there is a significant need for investigating the effects of treatment that is optimized for bilingual speakers with PPA. This stage 2 efficacy clinical trial seeks to establish the effects of culturally and linguistically tailored speech-language interventions administered to bilingual individuals with PPA.

The overall aim of the intervention component of this study is to establish the relationships between the bilingual experience (e.g., how often each language is used, how "strong" each language is) and treatment response of bilinguals with PPA. Specifically, the investigators will evaluate the benefits of tailored speech-language intervention administered in both languages to bilingual individuals with PPA (60 individuals will be recruited). The investigators will conduct an assessment before treatment, after treatment and at two follow-ups (6 and 12-months post-treatment) in both languages. When possible, a structural scan of the brain (magnetic resonance image) will be collected before treatment in order to identify if brain regions implicated in bilingualism are associated with response to treatment. In addition to the intervention described herein, 30 bilingual individuals with PPA will be recruited to complete behavioral cognitive-linguistic testing and will not receive intervention. Results will provide important knowledge about the neural mechanisms of language re-learning and will address how specific characteristics of bilingualism influence cognitive reserve and linguistic resilience in PPA.

ELIGIBILITY:
Inclusion Criteria:

* Meets diagnostic criteria for Primary Progressive Aphasia (PPA; Gorno-Tempini et al., 2011)
* Bilingual in Spanish and Catalan or bilingual in Spanish and English
* Different proficiency levels across languages are expected, any prior experience in both languages is acceptable
* Intervention study: Score of 15 or higher on the Mini-Mental State Examination
* Note that this project will also recruit individuals to participate in assessment only, for these individuals the following inclusion criteria applies: Score of 10 or higher on the Mini-Mental State Examination

Exclusion Criteria:

* Other central nervous system or medical diagnosis that can cause symptoms
* Other psychiatric diagnosis that can cause symptoms
* Significant, uncorrected visual or hearing impairment that would interfere with participation
* Prominent initial non-speech-language impairments (cognitive, behavioral, motoric)
* Intervention Study: Score of less than 15 on the Mini-Mental State Examination
* Note that this project will also recruit individuals to participate in assessment only, for these individuals the following inclusion criteria applies: Score of less than 10 on the Mini-Mental State Examination

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Percent correct intelligible words from trained/untrained scripts | Pre-phase 1, post-phase1/pre-phase 2 (4.5 weeks from treatment onset), post-phase 2 (9 weeks from treatment onset), 6 months and 1 year post-treatment
  Percent of intelligible, scripted words for trained scripts and untrained scripts
Percent correct spoken naming of trained/untrained nouns | Pre-phase 1, post-phase1/pre-phase 2 (4.5 weeks from treatment onset), post-phase 2 (9 weeks from treatment onset), 6 months and 1 year post-treatment
  Percent of correctly named trained pictured items and untrained pictured items

SECONDARY OUTCOMES:
Aphasia Impact Questionnaire (AIQ) | Pre-phase 1, Post-phase 2 (9 weeks from treatment onset)
  Patient reported outcome measure for use with people with aphasia comprising three sections: activities, participation and emotional state/wellbeing. Uses a 5 point pictorial rating scale. The minimum score is 0 (best) and the maximum is 4 (worst).
Connected Speech Features: Type-token ratio | Pre-phase 1, Post-phase1/pre-phase 2 (4.5 weeks from treatment onset), Post-phase 2 (9 weeks from treatment onset), 6 months and 1 year post-treatment
  Total number of unique words (types) divided by the total number of words (tokens) derived from connected speech samples (script topic probes, picture description, and personal narrative).
Connected Speech Features: Mean length of utterance | Pre-phase 1, Post-phase1/pre-phase 2 (4.5 weeks from treatment onset), Post-phase 2 (9 weeks from treatment onset), 6 months and 1 year post-treatment
  Average number of words produced per utterance derived from connected speech samples (script topic probes, picture description, and personal narrative).
Acoustic Features: Articulation Rate | Pre-phase 1, Post-phase1/pre-phase 2 (4.5 weeks from treatment onset), Post-phase 2 (9 weeks from treatment onset), 6 months and 1 year post-treatment
  Syllables per second of phonated time derived from connected speech samples (script topic probes, picture description, and personal narrative).
Acoustic Features: Speech-to-pause time | Pre-phase 1, Post-phase1/pre-phase 2 (4.5 weeks from treatment onset), Post-phase 2 (9 weeks from treatment onset), 6 months and 1 year post-treatment
  Phonated time divided by pause time in the sample derived from connected speech samples (script topic probes, picture description, and personal narrative).

OTHER OUTCOMES:
Post-treatment Communication Survey | Post-treatment (approximately 6-12 weeks after treatment onset)
  Survey characterizing perceived response to treatment. Scale scale options are as follows: "a lot worse", "worse", "somewhat worse", "unchanged", "somewhat better", "better", and "a lot better." There are seven levels with "a lot worse" being the lowest rating and "a lot better" being the best rating.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie M Grasso, Ph.D, Principal Investigator — University of Texas at Austin; Miguel Ángel Santos Santos, MD, PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (3):
- University of Texas at Austin, Austin, Texas, United States
- Spain (2):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Clínic de Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: Yes
Data generated from this project will be shared via peer reviewed journal publications as well as through national and international conferences. All peer-reviewed manuscripts will be made available via PubMed Central, in adherence to the NIH Public Access Policy. Intervention protocols, de-identified summary data, and software code/scripts used for data analysis will be made publicly available upon publication of trial results. De-identified data from individual participants may be made available to the scientific community with approved data use and sharing agreements between the University of Texas, Hospital Sant Pau, Hospital Clínic de Barcelona, and requesting institutions or entities, consistent with institution policy.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Intervention protocols, de-identified summary data, and software code/scripts used for data analysis will be made publicly available upon publication of trial results.
Access Criteria: De-identified data from individual participants may be made available to the scientific community with approved data use and sharing agreements between the University of Texas, Hospital Sant Pau, Hospital Clínic de Barcelona, and requesting institutions or entities, consistent with institution policy.

REFERENCES:
- [Background] Klimova B, Maresova P, Valis M, Hort J, Kuca K. Alzheimer's disease and language impairments: social intervention and medical treatment. Clin Interv Aging. 2015 Aug 27;10:1401-7. doi: 10.2147/CIA.S89714. eCollection 2015. PMID 26346123
- [Background] Szatloczki G, Hoffmann I, Vincze V, Kalman J, Pakaski M. Speaking in Alzheimer's Disease, is That an Early Sign? Importance of Changes in Language Abilities in Alzheimer's Disease. Front Aging Neurosci. 2015 Oct 20;7:195. doi: 10.3389/fnagi.2015.00195. eCollection 2015. PMID 26539107
- [Background] Mesulam MM. Slowly progressive aphasia without generalized dementia. Ann Neurol. 1982 Jun;11(6):592-8. doi: 10.1002/ana.410110607. PMID 7114808
- [Background] Montembeault M, Brambati SM, Gorno-Tempini ML, Migliaccio R. Clinical, Anatomical, and Pathological Features in the Three Variants of Primary Progressive Aphasia: A Review. Front Neurol. 2018 Aug 21;9:692. doi: 10.3389/fneur.2018.00692. eCollection 2018. PMID 30186225
- [Background] Gorno-Tempini ML, Hillis AE, Weintraub S, Kertesz A, Mendez M, Cappa SF, Ogar JM, Rohrer JD, Black S, Boeve BF, Manes F, Dronkers NF, Vandenberghe R, Rascovsky K, Patterson K, Miller BL, Knopman DS, Hodges JR, Mesulam MM, Grossman M. Classification of primary progressive aphasia and its variants. Neurology. 2011 Mar 15;76(11):1006-14. doi: 10.1212/WNL.0b013e31821103e6. Epub 2011 Feb 16. PMID 21325651
- [Background] Carthery-Goulart MT, da Silveira ADC, Machado TH, Mansur LL, Parente MAMP, Senaha MLH, Brucki SMD, Nitrini R. Nonpharmacological interventions for cognitive impairments following primary progressive aphasia: a systematic review of the literature. Dement Neuropsychol. 2013 Jan-Mar;7(1):122-131. doi: 10.1590/S1980-57642013DN70100018. PMID 29213828
- [Background] Bialystok E, Craik FI, Freedman M. Bilingualism as a protection against the onset of symptoms of dementia. Neuropsychologia. 2007 Jan 28;45(2):459-64. doi: 10.1016/j.neuropsychologia.2006.10.009. Epub 2006 Nov 27. PMID 17125807
- [Background] Alladi S, Bak TH, Shailaja M, Gollahalli D, Rajan A, Surampudi B, Hornberger M, Duggirala V, Chaudhuri JR, Kaul S. Bilingualism delays the onset of behavioral but not aphasic forms of frontotemporal dementia. Neuropsychologia. 2017 May;99:207-212. doi: 10.1016/j.neuropsychologia.2017.03.021. Epub 2017 Mar 18. PMID 28322905
- [Background] Alladi S, Bak TH, Duggirala V, Surampudi B, Shailaja M, Shukla AK, Chaudhuri JR, Kaul S. Bilingualism delays age at onset of dementia, independent of education and immigration status. Neurology. 2013 Nov 26;81(22):1938-44. doi: 10.1212/01.wnl.0000436620.33155.a4. Epub 2013 Nov 6. PMID 24198291
- [Background] de Leon J, Grasso SM, Welch A, Miller Z, Shwe W, Rabinovici GD, Miller BL, Henry ML, Gorno-Tempini ML. Effects of bilingualism on age at onset in two clinical Alzheimer's disease variants. Alzheimers Dement. 2020 Dec;16(12):1704-1713. doi: 10.1002/alz.12170. Epub 2020 Sep 3. PMID 32881346
- [Background] Costa AS, Jokel R, Villarejo A, Llamas-Velasco S, Domoto-Reilley K, Wojtala J, Reetz K, Machado A. Bilingualism in Primary Progressive Aphasia: A Retrospective Study on Clinical and Language Characteristics. Alzheimer Dis Assoc Disord. 2019 Jan-Mar;33(1):47-53. doi: 10.1097/WAD.0000000000000288. PMID 30640254
- [Background] Grasso SM, Pena ED, Kazemi N, Mirzapour H, Neupane R, Bonakdarpour B, Gorno-Tempini ML, Henry ML. Treatment for Anomia in Bilingual Speakers with Progressive Aphasia. Brain Sci. 2021 Oct 20;11(11):1371. doi: 10.3390/brainsci11111371. PMID 34827370
- [Background] Grasso SM, Shuster KM, Henry ML. Comparing the effects of clinician and caregiver-administered lexical retrieval training for progressive anomia. Neuropsychol Rehabil. 2019 Jul;29(6):866-895. doi: 10.1080/09602011.2017.1339358. Epub 2017 Jun 30. PMID 28662598
- [Background] Henry ML, Hubbard HI, Grasso SM, Mandelli ML, Wilson SM, Sathishkumar MT, Fridriksson J, Daigle W, Boxer AL, Miller BL, Gorno-Tempini ML. Retraining speech production and fluency in non-fluent/agrammatic primary progressive aphasia. Brain. 2018 Jun 1;141(6):1799-1814. doi: 10.1093/brain/awy101. PMID 29718131
- [Background] Henry ML, Hubbard HI, Grasso SM, Dial HR, Beeson PM, Miller BL, Gorno-Tempini ML. Treatment for Word Retrieval in Semantic and Logopenic Variants of Primary Progressive Aphasia: Immediate and Long-Term Outcomes. J Speech Lang Hear Res. 2019 Aug 15;62(8):2723-2749. doi: 10.1044/2018_JSLHR-L-18-0144. Epub 2019 Aug 7. PMID 31390290